CLINICAL TRIAL: NCT03991936
Title: Benefit of Placebo and Different Concentrations of Triamcinolone Acetonide in Nail Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1609017586
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Nail Psoriasis; Nail Diseases
Keywords: Nail Psoriasis; Nail Diseases; Triamcinolone acetonide; Triamcinolone
MeSH Terms: conditions — Nail Diseases | interventions — Saline Solution; Injections; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Placebo (Placebo Comparator): Participants receive an intralesional injection of 0.1-0.2 mL of normal saline in one psoriatic fingernail once per 6 weeks until 24 weeks.
  Interventions: Drug: Placebos
- Triamcinolone Acetonide 2.5 mg/mL (Experimental): Participants receive an intralesional injection of 0.1-0.2 mL of 2.5 mg/mL intralesional triamcinolone acetonide in one psoriatic fingernail once per 6 weeks until 24 weeks.
  Interventions: Drug: Triamcinolone Acetonide 2.5 mg/mL
- Triamcinolone Acetonide 5.0 mg/mL (Experimental): Participants receive an intralesional injection of 0.1-0.2 mL of 5.0 mg/mL intralesional triamcinolone acetonide in one psoriatic fingernail once per 6 weeks until 24 weeks.
  Interventions: Drug: Triamcinolone Acetonide 5.0 mg/mL
- Triamcinolone Acetonide 7.5 mg/mL (Experimental): Participants receive an intralesional injection of 0.1-0.2 mL of 7.5 mg/mL intralesional triamcinolone acetonide in one psoriatic fingernail once per 6 weeks until 24 weeks.
  Interventions: Drug: Triamcinolone Acetonide 7.5 mg/mL
- Triamcinolone Acetonide 10 mg/mL (Experimental): Participants receive an intralesional injection of 0.1-0.2 mL of 10 mg/mL intralesional triamcinolone acetonide in one psoriatic fingernail once per 6 weeks until 24 weeks.
  Interventions: Drug: Triamcinolone Acetonide 10 mg/mL

INTERVENTIONS:
Drug: Placebos — Normal saline intralesional injection
  Other Names: Saline solution for injection
  Arms: Placebo
Drug: Triamcinolone Acetonide 2.5 mg/mL — 2.5 mg/mL intralesional injection
  Other Names: Triamcinolone Injection; Kenalog 10 MG/ML Injectable Suspension
  Arms: Triamcinolone Acetonide 2.5 mg/mL
Drug: Triamcinolone Acetonide 5.0 mg/mL — 5.0 mg/mL intralesional injection
  Other Names: Triamcinolone Injection; Kenalog 10 MG/ML Injectable Suspension
  Arms: Triamcinolone Acetonide 5.0 mg/mL
Drug: Triamcinolone Acetonide 7.5 mg/mL — 7.5 mg/mL intralesional injection
  Other Names: Triamcinolone Injection; Kenalog 10 MG/ML Injectable Suspension
  Arms: Triamcinolone Acetonide 7.5 mg/mL
Drug: Triamcinolone Acetonide 10 mg/mL — 10 mg/mL intralesional injection
  Other Names: Triamcinolone Injection; Kenalog 10 MG/ML Injectable Suspension
  Arms: Triamcinolone Acetonide 10 mg/mL

SUMMARY:
This purpose of this study is to determine the lowest effective concentration of intralesional triamcinolone acetonide in the treatment of nail psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosed with nail psoriasis in at least 2 fingernails
* Willing to give written informed consent and able to adhere to procedures and visit schedules
* Must consent to having the fingernails photographed during the study period

Exclusion Criteria:

* Subject with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with study evaluations or optimal participation in the study. This is including, but not limited to: immunodeficiency, onychomycosis, any other nail condition other than psoriasis, allergy to triamcinolone acetonide, local anesthetic, normal saline, or any other material used for procedures
* Subject who has received radiation therapy, chemotherapy, and/or immunosuppressive drugs within 6 months of study, and/or oral corticosteroids for >1 month within the 6 months of study (exception: inhaled steroids)
* Subject known to have received treatment with investigational drugs or devices within 30 days prior to enrollment into this study
* Subject who is unwilling to abstain from any cosmetic nail treatments outside those provided by the study clinic, beyond basic nail trimming (i.e. no spa nail treatments, no nail polish use, no other topical prescription nail medication)
* Subject who is unwilling to abstain from any medical nail treatments on their nails other than the study intervention (i.e. topical steroids, anti-fungal creams) for the duration of the study intervention and for duration of the washout period (if applicable)
* Subject who is part of the staff personnel directly involved with this study or a family member of the investigational study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Lipner, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one location in the United States
Pre-assignment Details: A total of 11 participants passed screening and were randomized.
Units Other Than Participants: Fingernails
Period: Overall Study
Arm/Group | Placebo | Triamcinolone Acetonide 2.5 mg/mL | Triamcinolone Acetonide 5.0 mg/mL | Triamcinolone Acetonide 7.5 mg/mL | Triamcinolone Acetonide 10 mg/mL
Started | 11; 11 Fingernails | 11; 18 Fingernails | 11; 19 Fingernails | 11; 18 Fingernails | 11; 16 Fingernails
Completed | 10; 10 Fingernails | 10; 16 Fingernails | 10; 17 Fingernails | 10; 16 Fingernails | 10; 14 Fingernails
Not Completed | 1; 1 Fingernails | 1; 2 Fingernails | 1; 2 Fingernails | 1; 2 Fingernails | 1; 2 Fingernails
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Fingernails
Groups:
- All Participants: Participants receive an intralesional injection of 0.1-0.2 mL of 2.5 mg/mL, 5 mg/mL, 7.5 mg/mL or 10 mg/mL intralesional triamcinolone acetonide, or normal saline in one psoriatic fingernail once per 6 weeks until 24 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Number analyzed (Fingernails) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Nail Psoriasis Qualify of Life, as Measured by Development and Validation of Nail Psoriasis Quality [Mean (Full Range); unit: percentage of NPQ10 score] — The NPQ10 comprises 10 questions gauging the impact of nail psoriasis on daily activities. Each response is scored from 0 to 2, resulting in a total score between 0 and 20, where higher values indicate a more significant impact. The final scores are converted to percentages, reflecting the proportion of questions answered by the patient. The obtained score correlates proportionally with the level of functional difficulty experienced, with 0% indicating no impairment and 100% indicating the worst possible impairment.
  percentage of NPQ10 score | 7 [0 to 30]
Nail Psoriasis, as Measured by Nail Psoriasis Severity Index (NAPSI) [Mean (Full Range); unit: score on a scale] — The Nail Psoriasis Severity Index (NAPSI) is used to evaluate nail psoriasis. Scores range from 0 to 8 with 0 indicating no nail psoriasis and higher scores indicating worsening nail psoriasis Population: The Nail Psoriasis Severity Index (NAPSI) measure is provided for units, and the number of fingernails included in each arm varies. Data is presented per arm, and an additional "Total" row is added.
  score on a scale
    Triamcinolone acetonide 2.5 mg/mL: number analyzed (Fingernails) | 18
    Triamcinolone acetonide 2.5 mg/mL | 5.3 [3 to 8]
    Triamcinolone acetonide 5.0 mg/mL: number analyzed (Fingernails) | 19
    Triamcinolone acetonide 5.0 mg/mL | 4.76 [3 to 7]
    Triamcinolone acetonide 7.5 mg/mL: number analyzed (Fingernails) | 18
    Triamcinolone acetonide 7.5 mg/mL | 4.75 [3 to 7]
    Triamcinolone acetonide 10 mg/mL: number analyzed (Fingernails) | 16
    Triamcinolone acetonide 10 mg/mL | 5.0 [3 to 8]
    Placebo: number analyzed (Fingernails) | 11
    Placebo | 4.7 [3 to 6]
    Total | 4.9 [3 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Lowest Effective Concentration of Intralesional Triamcinolone Acetonide for Nail Psoriasis
Description: The most effective concentration of intralesional triamcinolone acetonide will be determined between 0 mg/mL, 2.5 mg/mL, 5.0 mg/mL, 7.5 mg/mL, and 10.0 mg/mL.
Time Frame: 24 weeks (end of study)
Population: Per protocol defined as participants completing 24-week follow-up visit
Measure: Number; unit: mg/mL
Units Other Than Participants: Fingernails
Groups:
- All Groups: Participants receive an intralesional injection of 0.1-0.2 mL of 2.5 mg/mL, 5 mg/mL, 7.5 mg/mL, or 10 mg/mL intralesional triamcinolone acetonide in one psoriatic fingernail once per 6 weeks until 24 weeks.
Arm/Group | All Groups
Number analyzed (Participants) | 10
Number analyzed (Fingernails) | 73
mg/mL | 2.5

2. Secondary Outcome: Change From Baseline in Nail Psoriasis, as Measured by Nail Psoriasis Severity Index (NAPSI)
Description: The Nail Psoriasis Severity Index (NAPSI) is used to evaluate nail psoriasis. Scores range from 0 to 8 with 0 indicating no nail psoriasis and higher scores indicating worsening nail psoriasis.
Time Frame: Baseline, 24 weeks (end of study)
Population: Per protocol population, defined as participants completing 24-week follow-up visit
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Fingernails
Arm/Group | Placebo | Triamcinolone Acetonide 2.5 mg/mL | Triamcinolone Acetonide 5.0 mg/mL | Triamcinolone Acetonide 7.5 mg/mL | Triamcinolone Acetonide 10 mg/mL
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Number analyzed (Fingernails) | 10 | 16 | 17 | 16 | 14
score on a scale | -0.96 [-1.81 to -0.11] | -3.96 [-4.64 to -3.27] | -2.96 [-3.62 to -2.31] | -3.53 [-4.2 to -2.85] | -3.93 [-4.62 to -3.24]
Statistical Analysis 1: Comparison: Placebo vs Triamcinolone Acetonide 2.5 mg/mL vs Triamcinolone Acetonide 5.0 mg/mL vs Triamcinolone Acetonide 7.5 mg/mL vs Triamcinolone Acetonide 10 mg/mL; The null hypothesis was that the change from baseline to 24 weeks in the Nail Psoriasis Severity Index (NAPSI) for the triamcinolone acetonide groups: 2.5 mg/mL, 5.0 mg/mL, 7.5 mg/mL, and 10 mg/mL would be no different than the change from baseline to 24 weeks for the placebo group; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical analysis was p = 0.05; Mean Difference (Net) = -2.635

3. Secondary Outcome: Change From Baseline in Nail Psoriasis Qualify of Life, as Measured by Development and Validation of Nail Psoriasis Quality of Life Scale (NPQ10)
Description: The NPQ10 comprises 10 questions gauging the impact of nail psoriasis on daily activities. Each response is scored from 0 to 2, resulting in a total score between 0 and 20, where higher values indicate a more significant impact. The final scores are converted to percentages, reflecting the proportion of questions answered by the patient. The obtained score correlates proportionally with the level of functional difficulty experienced, with 0% indicating no impairment and 100% indicating the worst possible impairment.
Time Frame: Baseline, 24 weeks (end of study)
Population: Per protocol population, defined as participants completing the 24-week follow-up visit.
Measure: Mean (Full Range); unit: percentage of NPQ10 score
Groups:
- All Groups: Participants receive an intralesional injection of 0.1-0.2 mL of normal saline, 2.5 mg/m, 5 mg/ml, 7.5 mg/ml, or 10 mg/ml in one psoriatic fingernail once per 6 weeks until 24 weeks.
  All groups.
Arm/Group | All Groups
Number analyzed (Participants) | 10
percentage of NPQ10 score | 4.5 [0 to 15]

4. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: Adverse events will only include those that are determined to be related to the study drug.
Time Frame: 24 weeks (end of study)
Measure: Count of Participants; unit: Participants
Groups:
- Triamcinolone Acetonide 2.5 mg/mL: Participants receive an intralesional injection of 0.1-0.2 mL of 2.5 mg/mL, once per 6 weeks until 24 weeks.
- Triamcinolone Acetonide 5.0 mg/mL: Participants receive an intralesional injection of 0.1-0.2 mL of 5.0 mg/mL, once per 6 weeks until 24 weeks.
- Triamcinolone Acetonide 7.5 mg/mL: Participants receive an intralesional injection of 0.1-0.2 mL of 7.5 mg/mL, once per 6 weeks until 24 weeks.
- Triamcinolone Acetonide 10 mg/mL: Participants receive an intralesional injection of 0.1-0.2 mL of 10 mg/mL, once per 6 weeks until 24 weeks.
- Placebo: Participants receive an intralesional injection of 0.1-0.2 mL of normal saline, once per 6 weeks until 24 weeks.
Arm/Group | Triamcinolone Acetonide 2.5 mg/mL | Triamcinolone Acetonide 5.0 mg/mL | Triamcinolone Acetonide 7.5 mg/mL | Triamcinolone Acetonide 10 mg/mL | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 3 | 4 | 7 | 8 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events are reported using fingernails as unit. Adverse events were recorded for 10 subjects because one participant was lost to follow-up.
Arm/Group | Placebo | Triamcinolone Acetonide 2.5 mg/mL | Triamcinolone Acetonide 5.0 mg/mL | Triamcinolone Acetonide 7.5 mg/mL | Triamcinolone Acetonide 10 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 4/10 | 6/10 | 10/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Triamcinolone Acetonide 2.5 mg/mL (N=10) | Triamcinolone Acetonide 5.0 mg/mL (N=10) | Triamcinolone Acetonide 7.5 mg/mL (N=10) | Triamcinolone Acetonide 10 mg/mL (N=10)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 1 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 3/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 0/17 in the TAC 5.0 mg/mL group 3/16 in the TAC 7.5 mg/mL group 1/14 in the TAC 10 mg/mL group
Subungual hematoma (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 1/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 1/17 in the TAC 5.0 mg/mL group 1/16 in the TAC 7.5 mg/mL group 0/14 in the TAC 10 mg/mL group
Cuticle retraction (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 4 | 4 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 1/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 3/17 in the TAC 5.0 mg/mL group 6/16 in the TAC 7.5 mg/mL group 6/14 in the TAC 10 mg/mL group
Longitudinal groove (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 0/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 0/17 in the TAC 5.0 mg/mL group 2/16 in the TAC 7.5 mg/mL group 0/14 in the TAC 10 mg/mL group
Beau's line(s) (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 1/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 1/17 in the TAC 5.0 mg/mL group 1/16 in the TAC 7.5 mg/mL group 1/14 in the TAC 10 mg/mL group
Erythronychia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 2 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 1/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 1/17 in the TAC 5.0 mg/mL group 2/16 in the TAC 7.5 mg/mL group 2/14 in the TAC 10 mg/mL group
Nail plate split (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 0/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 0/17 in the TAC 5.0 mg/mL group 0/16 in the TAC 7.5 mg/mL group 1/14 in the TAC 10 mg/mL group
Nail plate concavity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 — Units (fingernails) affected/at risk: 0/10 in the Placebo group 0/16 in the triamcinolone acetonide (TAC) 2.5 mg/mL group 0/17 in the TAC 5.0 mg/mL group 0/16 in the TAC 7.5 mg/mL group 1/14 in the TAC 10 mg/mL group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03991936/Prot_SAP_000.pdf